CLINICAL TRIAL: NCT00684034
Title: Redox State in the Course of Chronic Renal Insufficiency and Hemodialysis: Implications in Morbimortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2007-A01179-44; 2007-38
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Renal Insufficiency
Keywords: Redox state in the course of chronic renal insufficiency and hemodialysis.
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Volunteer healthy
  Interventions: Other: Sampling of blood
- 2 (Other): Patient dialysis patient
  Interventions: Other: Sampling of blood
- 3 (Other): Not dialysed chronic renal insufficient patient
  Interventions: Other: Sampling of blood

INTERVENTIONS:
Other: Sampling of blood — A sampling of blood will be made
  Arms: 1
Other: Sampling of blood — A sampling of bood will be made before the dialysis
  Arms: 2
Other: Sampling of blood — A sampling of blood will be made.
  Arms: 3

SUMMARY:
The influence of hemodialysis on oxidative stress, endothelial activation, inflammation and on the redox state of lymphocytes should be clarified as well as the putative relationships between all these parameters.

DETAILED DESCRIPTION:
Up to now, no anti-oxydative treatment has been able to reduce the mortality of the patients with Kidney Failure. Thus it is necessary to have a better knowledge of oxydative stress mechanisms in patients with KF in order to find more efficacious treatments. The influence of hemodialysis upon oxidative stress is not well known.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 80 years old man or woman dialysing at least 3 times a week for at least 6 months and having no residual renal function
* Rate of haemoglobin > 11 g / dl
* Clinically stable patient that is having had no considerable event (cardiovascular problem, infection, surgical operation) with the exception of angioplasty of fistula or prosthesis vascular, in the previous 3 months the entrance to the study
* Patient capable of understanding and of following the essay, in particular knowing how to read the note of information.

Exclusion Criteria:

* Pregnant woman
* Treatment by corticoids or immunosuppresseurs
* hemopathy sly
* chronic cancer or infection in evolution
* Cardiovascular event (infarct, unstable angor, coronary bypasses, confusions of the rhythm, AVC, amputation) or infectious (blood-poisoning, pneumopathie, meningitis) or surgical operation in the previous 3 months the inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2008-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
This study should allow to clarify the redox state some plasma by quantification of thiols membranous on the surface of lymphocytes at the hemodialysis and insufficient renal chronic not dialysed patients. | 48 months

SECONDARY OUTCOMES:
This study should allow to estimate in a forward-looking longitudinal plan the possible involvement of the parameters of the redox state and the morbidity and the cardiovascular and global mortality in 2 years in 2 studied populations. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand DUSSOL, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Hopital de la Conception- Service de Néphrologie et de transplantation rénale, Marseille, France